CLINICAL TRIAL: NCT02113592
Title: Collaborative Care for Chronic Pain in Primary Care
Brief Title: Pain Program for Active Coping & Training
Acronym: PPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Duke University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00004169; UH3NS088731 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-14 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-04

CONDITIONS: Chronic Non-malignant Pain
Keywords: Pain management; Opioid use; Pragmatic; Collaborative care; Primary care
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interdisciplinary pain program (Experimental): Interdisciplinary pain program, which includes behavioral health, nurse case management, physical therapy, and pharmacy embedded in primary care.
  Interventions: Behavioral: Interdisciplinary pain program
- Treatment as usual (No Intervention): Patients in this arm will receive care as usual and utilize services as they currently exist in the health plan system.

INTERVENTIONS:
Behavioral: Interdisciplinary pain program — Interdisciplinary pain program, which includes behavioral health, nurse case management, physical therapy, and pharmacy embedded in primary care.
  Arms: Interdisciplinary pain program

SUMMARY:
The overall aim of this study is to adopt an integrative rehabilitation approach for helping patients adopt self-management skills for managing chronic pain, limiting use of opioid medications, and identifying exacerbating factors amenable to treatment (e.g., depression, sleep problems) that is feasible and sustainable within the primary care setting.

DETAILED DESCRIPTION:
Pain is a common and very costly public health problem. Common chronic pain conditions are expensive and pervasive, affecting at least 116 million American adults at an annual cost of $560 billion in direct medical treatment costs and lost productivity, and disproportionally affect vulnerable populations. Pain is the primary reason patients seek medical care and, as the first point of contact, primary care providers (PCPs) deliver the majority of that care. Unfortunately, PCPs face many challenges in managing these patients' care and often have little specific training in pain medicine. Yet with proper system support, PCPs are in the best position to coordinate pain management longitudinally. While pharmacotherapy is the predominant treatment approach for many PCPs, this limits the patient's role to taking medication, and he or she can become a passive recipient of care-leading to poor outcomes, potential overmedication, and possible disillusionment with the medical system. Further, increases in opiate prescribing for pain treatment-amidst increasing awareness of adverse outcomes, including addiction-and limited efficacy suggest the importance of broader treatment approaches that focus on patients' improvement of functioning. Although opiates may reduce pain symptoms while prescribed, patients are unlikely to experience significant and sustained improvements without the use of other nonpharmacologic pain management approaches. Medical management of patients with persistent pain and complex problems is often fragmented, which leads patients to seek a wide variety of primary and specialty care services in an effort to manage their pain and related conditions. Such fragmented care leads to poorer outcomes and significantly increases health care costs as patients often receive unneeded diagnostic and medical procedures. While research has identified evidence-based multidisciplinary behavioral treatment approaches that are effective for such patients and can even prevent the disability associated with persistent pain when offered earlier in the course of care, these interventions are rarely available in everyday practice settings and will require data from pragmatic clinical trials to change the care paradigm.

To address these issues, we are conducting a large-scale, mixed-methods, cluster-randomized pragmatic clinical trial throughout three regions of Kaiser Permanente - Northwest, Georgia, and Hawaii. This trial will evaluate the integration of multidisciplinary services within the primary care environment as compared to usual care in these settings. This project embeds an intervention into everyday clinical practice flow utilizing assessment measures and intervention staff directly from the clinical care system rather than utilizing a research-developed and administered structure. The intervention is an integrated, interdisciplinary program that guides all pain-related care for intervention patients. This study compares this primary care-based intervention to usual care using systematic, clinic-based assessments. The trial will include up to 1,000 patients and 500 primary care providers (half of each receiving active treatment) with intervention care being delivered by behavioral specialists, nurses, physical therapists, pharmacists, and other affiliated staff. Patients include those selected by their primary care providers who have non-malignant chronic pain (pain persisting for ≥ 3 months) and who are on long-term opiate therapy for the treatment of their condition. This intervention brings together elements often available in health plans but organized in a less integrated fashion, and it will ensure flexibility in implementation to best fit individual clinic environments and the needs of chronic pain patients on long-term opiate therapy.

ELIGIBILITY:
Patient inclusion criteria are:

1. Adult (18 years of age or older) Kaiser Permanente (KP) health plan members from the KP Northwest, KP Georgia, and KP Hawaii regions who receive their primary care services from participating primary care providers
2. Kaiser Permanente health plan membership of at least 180 days duration
3. Long term opioid use defined by: 90+ day supply of short acting opioid spanning at least 120 days or 2 or more long acting opioid dispense in the past 180 days
4. Pain diagnosis within the past year (based on ICD-9 or ICD-10 diagnostic codes)
5. English speaking

Patient exclusion criteria are:

1. Currently enrolled in intensive addiction medicine services or evidence of active substance dependence
2. Cognitive impairment severe enough to preclude patient's participation in a behavioral/lifestyle change program
3. Current malignant cancer diagnosis
4. Having received hospice or other end-of-life palliative care within past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente Center for Health Research, Atlanta, Georgia
  - Kaiser Permanente Center for Health Research, Honolulu, Hawaii
  - Kaiser Permanente Center for Health Research, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith DH, O'Keeffe-Rosetti M, Leo MC, Mayhew M, Benes L, Bonifay A, Deyo RA, Elder CR, Keefe FJ, McMullen C, Owen-Smith A, Trinacty CM, Vollmer WM, DeBar L. Economic Evaluation: A Randomized Pragmatic Trial of a Primary Care-based Cognitive Behavioral Intervention for Adults Receiving Long-term Opioids for Chronic Pain. Med Care. 2022 Jun 1;60(6):423-431. doi: 10.1097/MLR.0000000000001713. Epub 2022 Mar 30. PMID 35352703
- [Result] DeBar L, Mayhew M, Benes L, Bonifay A, Deyo RA, Elder CR, Keefe FJ, Leo MC, McMullen C, Owen-Smith A, Smith DH, Trinacty CM, Vollmer WM. A Primary Care-Based Cognitive Behavioral Therapy Intervention for Long-Term Opioid Users With Chronic Pain : A Randomized Pragmatic Trial. Ann Intern Med. 2022 Jan;175(1):46-55. doi: 10.7326/M21-1436. Epub 2021 Nov 2. PMID 34724405
- [Derived] Mayhew M, Leo MC, Vollmer WM, DeBar LL, Kiernan M. Interactive group-based orientation sessions: A method to improve adherence and retention in pragmatic clinical trials. Contemp Clin Trials Commun. 2020 Jan 21;17:100527. doi: 10.1016/j.conctc.2020.100527. eCollection 2020 Mar. PMID 32083219
- [Derived] Owen-Smith A, Mayhew M, Leo MC, Varga A, Benes L, Bonifay A, DeBar L. Automating Collection of Pain-Related Patient-Reported Outcomes to Enhance Clinical Care and Research. J Gen Intern Med. 2018 May;33(Suppl 1):31-37. doi: 10.1007/s11606-018-4326-9. PMID 29633139
- [Derived] DeBar L, Benes L, Bonifay A, Deyo RA, Elder CR, Keefe FJ, Leo MC, McMullen C, Mayhew M, Owen-Smith A, Smith DH, Trinacty CM, Vollmer WM. Interdisciplinary team-based care for patients with chronic pain on long-term opioid treatment in primary care (PPACT) - Protocol for a pragmatic cluster randomized trial. Contemp Clin Trials. 2018 Apr;67:91-99. doi: 10.1016/j.cct.2018.02.015. Epub 2018 Mar 6. PMID 29522897
- [Derived] Johnson KE, Neta G, Dember LM, Coronado GD, Suls J, Chambers DA, Rundell S, Smith DH, Liu B, Taplin S, Stoney CM, Farrell MM, Glasgow RE. Use of PRECIS ratings in the National Institutes of Health (NIH) Health Care Systems Research Collaboratory. Trials. 2016 Jan 16;17:32. doi: 10.1186/s13063-016-1158-y. PMID 26772801

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Primary care provider cluster
Groups:
- Cognitive Behavioral Therapy (CBT) Intervention: Cognitive behavioral therapy (CBT) intervention teaching pain self-management skills in 12 weekly, 90-minute groups delivered by an interdisciplinary team of a behavioral health specialist, nurse care manager, physical therapist, and pharmacist, embedded in primary care.
- Usual Care: Patients in this arm receive care as usual and can utilize any pharmacologic and/or nonpharmacologic treatments available to them in their health care system without restriction.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Started | 433; 53 Primary care provider cluster | 417; 53 Primary care provider cluster
Completed | 414; 53 Primary care provider cluster | 402; 53 Primary care provider cluster
Not Completed | 19; 0 Primary care provider cluster | 15; 0 Primary care provider cluster

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care | Total
Number analyzed (Participants) | 433 | 417 | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.9) | 59.2 (12.4) | 60.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 286 | 573
  Male | 146 | 131 | 277
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic ethnicity | 16 | 12 | 28
  White (race) | 334 | 317 | 651
  Black or African American (race) | 55 | 55 | 110
  Other (race) | 44 | 45 | 89
Region of Enrollment [Number; unit: participants]
  United States | 433 | 417 | 850
Average daily dose of opioids [Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents (MME)] | 28.5 [16.0 to 53.2] | 30.8 [16.0 to 75.1] | 29.6 [16.0 to 62.0]

OUTCOME MEASURES:

1. Primary Outcome: Pain Impact Assessed Using the 4-Item Version of Brief Pain Inventory-Short Form ("PEGS")
Description: Reliable and valid tool that measures patients' pain intensity and functional interference. The primary outcome of pain impact is assessed with the 4-item PEGS scale, a composite of pain intensity, and interference with enjoyment of life, general activity, and sleep (range, 0-10, higher score = worse pain impact).
Time Frame: Collected every 3 months for 1 year
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 414 | 402
score on a scale
  Baseline | 6.485 [6.290 to 6.681] | 6.645 [6.447 to 6.843]
  3-Month Follow-Up | 5.486 [5.272 to 5.699] | 6.210 [5.994 to 6.426]
  6-Month Follow-Up | 5.516 [5.316 to 5.715] | 6.197 [5.994 to 6.399]
  9-Month Follow-up | 5.546 [5.342 to 5.750] | 6.183 [5.976 to 6.390]
  12-Month Follow-Up | 5.576 [5.349 to 5.803] | 6.170 [5.940 to 6.400]

2. Secondary Outcome: Pain-related Disability
Description: Pain-related disability will be assessed using the 24-item Roland Morris Disability Questionnaire (range, 0-1, higher score = worse function)
Time Frame: Collected every 3 months for 1 year
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 414 | 402
score on a scale
  Baseline | 0.672 [0.652 to 0.691] | 0.692 [0.672 to 0.711]
  3-Month Follow-Up | 0.612 [0.591 to 0.633] | 0.675 [0.654 to 0.696]
  6-Month Follow-Up | 0.609 [0.590 to 0.629] | 0.678 [0.658 to 0.698]
  9-Month Follow-Up | 0.607 [0.586 to 0.627] | 0.681 [0.660 to 0.701]
  12-Month Follow-Up | 0.604 [0.581 to 0.626] | 0.683 [0.661 to 0.706]

3. Secondary Outcome: Average Daily Dose of Opioids
Description: Average daily dose of opioids per 3-month quarter measured in morphine milligram equivalents (MME)
Time Frame: Collected every 3 months for 1 year
Measure: Mean (95% Confidence Interval); unit: MME/day
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 414 | 402
MME/day
  Baseline | 47.458 [40.647 to 54.269] | 55.252 [48.333 to 62.171]
  3-Month Follow-Up | 46.641 [39.610 to 53.627] | 56.695 [49.556 to 63.834]
  6-Month Follow-Up | 45.606 [38.574 to 52.638] | 55.563 [48.421 to 62.704]
  9-Month Follow-Up | 44.571 [37.396 to 51.745] | 54.430 [47.142 to 61.719]
  12-Month Follow-Up | 43.536 [36.085 to 50.986] | 53.298 [45.725 to 60.871]

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with health care services will be assessed using two distinct items:
  * [Satisfaction with primary care services]: In the past 3 months, how satisfied have you been with your primary care services? (1, Very dissatisfied; 2, Mildly dissatisfied; 3, Indifferent; 4, Mostly satisfied; 5, Very satisfied)
  * [Satisfaction with pain services]: In the past 3 months, how satisfied have you been with the pain services you have received? (1, Very dissatisfied; 2, Mildly dissatisfied; 3, Indifferent; 4, Mostly satisfied; 5, Very satisfied)
  Each item is scored individually; (range=1-5, higher score = greater satisfaction)
Time Frame: Collected at baseline and 6 months (post-treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 414 | 402
score on a scale
  Satisfaction with primary care services (Baseline) | 4.263 [4.162 to 4.365] | 4.237 [4.134 to 4.339]
  Satisfaction with primary care services (Post-Treatment) | 4.240 [4.115 to 4.365] | 3.984 [3.856 to 4.112]
  Satisfaction with pain services (Baseline) | 3.658 [3.540 to 3.776] | 3.581 [3.461 to 3.700]
  Satisfaction with pain services (Post-Treatment) | 4.080 [3.954 to 4.205] | 3.667 [3.538 to 3.796]

5. Secondary Outcome: Health Care Costs
Description: Costs were measured based on patient utilization of health care services and all prescription/medication costs. The costs of health care encounters during the 1-year follow-up were estimated using the standardized relative resource cost algorithm (SRRCA).
  Pain-related health care costs were based on the pain-related health care encounters identified using diagnostic and procedure coding.
Time Frame: Collected for 1 year post-randomization
Measure: Mean (95% Confidence Interval); unit: Dollars
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 412 | 402
Dollars
  Total Health Care Costs | 21,372 [18,114 to 24,630] | 25,648 [22,350 to 28,946]
  Total Pain-Related Health Care Costs | 9,395 [7,216 to 11,574] | 11,343 [9,137 to 13,549]

6. Secondary Outcome: Count of Health Care Encounters by Type (Health Care Utilization)
Description: Total Ambulatory Encounters includes encounters in the following health care service categories: Primary care; Physical therapy; Pain clinic; Other specialty medical care; Mental health; Complementary and alternative medicine; ED, urgent care, and observation beds; Hospital ambulatory visits; Same day surgeries; and Home health.
  Total Pain-Related Ambulatory Encounters are a subset of Total Ambulatory Encounters and were identified using CPT, HCPCS, and ICD-9-PCS or ICD-10-PCS codes
Time Frame: Collected for 1 year post-randomization
Measure: Mean (95% Confidence Interval); unit: Health care encounters
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 412 | 402
Health care encounters
  Total Ambulatory Encounters | 20.85 [19.40 to 22.41] | 21.59 [20.07 to 23.22]
  Total Pain-Related Ambulatory Encounters | 10.42 [9.62 to 11.28] | 10.11 [9.33 to 10.96]
  Telephone or Email Encounters | 24.04 [22.57 to 25.60] | 23.18 [21.75 to 24.71]
  Inpatient Hospital Encounters | 0.22 [0.17 to 0.28] | 0.28 [0.22 to 0.36]

7. Secondary Outcome: Inpatient Hospital Days (Health Care Utilization)
Description: Inpatient hospital days is the average number of days that patients stayed in hospital (total number of days spent by inpatients during the 1 year post-randomization divided by the total number of inpatient admissions)
Time Frame: Collected for 1 year post-randomization
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 412 | 402
Days | 0.86 [0.59 to 1.26] | 0.22 [0.13 to 0.39]

8. Secondary Outcome: Total Pharmacy Dispenses (Health Care Utilization)
Description: Total Pharmacy Dispenses is a count of the unique medication prescriptions dispensed.
Time Frame: Collected for 1 year post-randomization
Measure: Mean (95% Confidence Interval); unit: Prescriptions dispensed
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
Number analyzed (Participants) | 412 | 402
Prescriptions dispensed | 50.45 [48.53 to 52.44] | 52.22 [50.21 to 54.30]

ADVERSE EVENTS:
Time Frame: Participants were monitored for serious adverse events during the one-year period of study participation.
Description: The only adverse events monitored were serious adverse events, defined as hospitalizations and deaths, assessed systematically from electronic health record data. Assessments were conducted every 6 months throughout the study and reviewed by an independent monitor. For deaths, chart abstraction determined relatedness.
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/433 | 8/417
Serious Adverse Events (participants affected / at risk) | 94/433 | 112/417
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) Intervention (N=433) | Usual Care (N=417)
Hospitalization (General disorders) | 94 (116) | 112 (171) — All hospitalizations were unrelated to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02113592/Prot_SAP_000.pdf